CLINICAL TRIAL: NCT01436526
Title: Single-dose, Open-label, Randomized, 2-way Crossover Pivotal Bioequivalence Study of 2x5 mg Tablets Rivaroxaban Versus 1x10 mg Tablet Rivaroxaban Under Fasted Condition in Healthy Subjects
Brief Title: Bioequivalence Study in Healthy Subjects, 2*5 mg Tablets Rivaroxaban Versus 1*10 mg Tablet Rivaroxaban
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 14588; 2009-013032-20 (EudraCT Number)
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Therapeutic Equivalency
Keywords: Bioequivalence
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) first 2*5 mg, then 1*10 mg (Experimental): Single oral dose of rivaroxaban administered under fasting conditions 2*5 mg tablet in first intervention period and 1*10 mg tablet in second intervention period (after washout period)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Rivaroxaban (Xarelto, BAY59-7939) first 1*10 mg, then 2*5 mg (Experimental): Single oral dose of rivaroxaban administered under fasting conditions 1*10 mg tablet in first intervention period and 2*5 mg tablet in second intervention period (after washout period)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Single oral dose of rivaroxaban administered under fasting conditions 2*5 mg tablet in first intervention period and 1*10 mg tablet in second intervention period (after washout period)
  Arms: Rivaroxaban (Xarelto, BAY59-7939) first 2*5 mg, then 1*10 mg
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Single oral dose of rivaroxaban administered under fasting conditions 1*10 mg tablet in first intervention period and 2*5 mg tablet in second intervention period (after washout period)
  Arms: Rivaroxaban (Xarelto, BAY59-7939) first 1*10 mg, then 2*5 mg

SUMMARY:
The drug investigated in this study is Rivaroxaban, a novel, once-daily, oral anticoagulant for the prevention (prophylaxis) of deep vein thrombosis (DVT) which may lead to a pulmonary embolism (PE) in people undergoing knee or hip replacement surgery.

The purpose of this study is to establish bioequivalence of 2 immediate-release tablet treatments with Rivaroxaban: 2*5 mg tablets and 1*10 mg tablet will be given to healthy volunteers under fasting conditions; they will be administered as single oral doses in 2 periods. Both periods will be separated by a 7-day washout phase. Thus, the bioequivalence represents the primary study objective. As a secondary objective, this treatment will be assessed in terms of safety and tolerability.

Bioequivalence will be evaluated and verified on the basis of pharmacokinetic data. Blood samples of the volunteers will be taken at specific points in time; these samples will be analyzed using various statistical methods to establish pharmacokinetic characteristics required to compare the 2 treatments. The planned treatments with Rivaroxaban will be considered bioequivalent if specific criteria defined in the study protocol are met.

The study will be conducted in one center in Germany. 28 subjects meeting the inclusion criteria will participate. They will be treated according to a single-dose, randomized, 2-way cross-over, non-placebo-controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* 18 to 45 years of age
* Body mass index (BMI) between 18 and 30 kg/m2

Exclusion Criteria:

* Conspicuous findings (medical history, screening)
* History of relevant diseases (internal organs, central nervous system or other organs)
* Medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Febrile illness within 1 week before the start of the study
* History of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Hypersensitivity to the investigational drug, the control agent and/or to inactive constituents
* Known coagulation disorders, known disorders with increased bleeding risk, known sensitivity to common causes of bleeding

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants (part.) recruited by CRS Clinical-Research-Services Moenchengladbach GmbH, Hindenburgstrasse 304 - 306, 41061 Moenchengladbach, Germany. 28 part. were planned to be enrolled.
Pre-assignment Details: 37 participants screened; 9 participants were screening failures; 28 participants were included in the study. Safety analysis: 27 individuals were analyzed in the group with 2*5mg, 27 individuals were analyzed in the group with 1*10mg.
Period: Period 1
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) First 2*5 mg, Then 1*10 mg | Rivaroxaban (Xarelto, BAY59-7939) First 1*10 mg, Then 2*5 mg
Started | 14 | 14
Participants Received Treatment | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) First 2*5 mg, Then 1*10 mg | Rivaroxaban (Xarelto, BAY59-7939) First 1*10 mg, Then 2*5 mg
Started | 13 (1 participant withdrew his consent after completing the first period.) | 13 (1 participant withdrew his consent after completing the first period.)
Participants Received Treatment | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rivaroxaban (Xarelto, BAY59-7939) First 2*5 mg , Then 1*10 mg: Single oral dose of rivaroxaban administered under fasting conditions 2*5 mg tablet in first intervention period and 1*10 mg tablet in second intervention period (after washout period)
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) First 2*5 mg , Then 1*10 mg | Rivaroxaban (Xarelto, BAY59-7939) First 1*10 mg, Then 2*5 mg | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.6 (5.8) | 31.3 (10.5) | 31.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity After Single Dose (AUC) Incl. Bioequivalence (BE) Evaluation
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample (AUC is defined as area under the concentration vs. time curve from zero to infinity after single (first) dose).
Time Frame: 0 min, 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 15 hours, 24 hours, 36 hours, 48 hours and 72 hours post administration
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/L
Groups:
- Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg: Single oral dose of 2*5 mg rivaroxaban tablet administered under fasting conditions
- Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg: Single oral dose of 1*10 mg rivaroxaban tablets administered under fasting conditions
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
µg*hr/L | 1374 (29.3) | 1268 (30.7)
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg vs Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg; Test type: Non-Inferiority or Equivalence — Using an estimated intra-subject coefficient of variation of less than 20% for AUC and Cmax, and a level of significance of 5%, a sample size of 25 completers was considered sufficient to conclude bioequivalence between 2*5 mg and 1*10 mg rivaroxaban with 90% power, if the 2 treatment means differed by 5%; p = 0.0438, ANOVA; LS-Mean Ratio, Percent = 108.35, 90% CI [101.59 to 115.57]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Last Quantifiable Concentration [AUC (0-tn)] Incl. Bioequivalence (BE) Evaluation
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; [AUC (0-tn)] is defined as AUC from time 0 to the last data point above the Lower Limit of Quantification.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/L
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
µg*hr/L | 1354 (29.8) | 1252 (31.6)
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg vs Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0514, ANOVA; LS-Mean Ratio, Percent = 108.19, 90% CI [101.31 to 115.54]

3. Primary Outcome: Maximum Observed Drug Concentration in Plasma After Single Dose Administration (Cmax) Incl. Bioequivalence (BE) Evaluation
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
µg/L | 179.8 (31.1) | 161.1 (38.7)
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg vs Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0685, ANOVA; LS-Mean Ratio, Percent = 111.64, 90% CI [101.14 to 123.23]

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Divided by Dose Per kg Body Weight (AUCnorm)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; AUCnorm is defined as AUC divided by dose per kg body weight.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg*hr/L
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
kg*hr/L | 10.79 (33.0) | 9.957 (36.4)

5. Secondary Outcome: Maximum Observed Drug Concentration in Plasma After Single Dose Administration Divided by Dose Per kg Body Weight (Cmax, Norm)
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; Cmax,norm is defined as Cmax divided by dose (mg) per kg body weight.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg/L
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
kg/L | 1.412 (35.3) | 1.265 (46.0)

6. Secondary Outcome: Mean Residence Time (MRT)
Description: The mean residence time is the average time that the molecules introduced into the body stay in the body.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
hr | 8.874 (22.0) | 9.284 (28.2)

7. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma After Single Dose (Tmax)
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Median (Full Range); unit: hr
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
hr | 2.50 [0.75 to 3.00] | 2.50 [0.75 to 4.00]

8. Secondary Outcome: Half-life Associated With the Terminal Slope (t½)
Description: Half-life refers to the elimination of the drug, i.e. the time it takes for the blood plasma concentration to reach half the concentration in the terminal phase of elimination.
Time Frame: as for outcome 1
Population: N=26 valid for pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 2*5 mg | Rivaroxaban (Xarelto, BAY59-7939) 1*10 mg
Number analyzed (Participants) | 26 | 26
hr | 8.932 (48.6) | 8.721 (55.7)

ADVERSE EVENTS:
Groups:
- Rivaroxaban 2*5 mg (Xarelto, BAY59-7939): Single oral dose of 2*5 mg rivaroxaban tablets administered under fasting conditions
- Rivaroxaban 1*10 mg (Xarelto, BAY59-7939): Single oral dose of 1*10 mg rivaroxaban tablet administered under fasting conditions
Arm/Group | Rivaroxaban 2*5 mg (Xarelto, BAY59-7939) | Rivaroxaban 1*10 mg (Xarelto, BAY59-7939)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 6/27 | 6/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 2*5 mg (Xarelto, BAY59-7939) (N=27) | Rivaroxaban 1*10 mg (Xarelto, BAY59-7939) (N=27)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood amylase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Glutamate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any disclosure of study results by the Principal Investigator or investigators has to be in agreement with the sponsor.